CLINICAL TRIAL: NCT01919957
Title: Etude de la mémoire Avant et après Chirurgie d'Une épilepsie Partielle pharmacorésistante : Bases Neurobiologiques, Applications Cliniques
Brief Title: Episodic Memory Before and After Surgery in Drug-resistant Partial Epilepsies
Acronym: MemO-Epi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C12-11; 2013-A00343-42 (Registry Identifier: C12-11)
Record Dates: First submitted 2013-07-01; First posted 2013-08-09 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy, Unspecified, Pharmacologically Resistant; Memory Impairment
Keywords: epilepsy; surgery; functional MRI; memory outcome
MeSH Terms: conditions — Epilepsy; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- memory outcome (No Intervention)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study has two purposes: firstly, a better understanding of the neurobiological processes underlying episodic memory and, secondly, the development of useful clinical applications for epileptic patients, in particular the prediction of postoperative memory deficits and the development of cognitive remediation therapies.

Memory performances during a fMRI experiment will be assessed in controls and epileptic patients before and after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with drug-resistant epilepsy
* Age of 18 years or more
* Follow-up in the epilepsy unit at Pitié-Salpêtrière Hospital
* Before or after the presurgical evaluation unit including a video-EEG monitoring, a structural brain imaging and a full neuropsychological assessment
* Covered by a social security system
* Signing of consent form

Exclusion Criteria:

* Persons under guardianship, curatorship or any other administrative or judicial deprivation of rights and freedom
* Refusal to consent form
* Contraindications to MRI
* Pregnancy
* Refusal to be informed in the case of detection of an abnormality during the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Measure of successfull encoding | 8 years
  Our goal is to define correlation between the measure of successfull object encoding trials (especially for binding) and the beta value activation in fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Dupont, MD, PhD, Principal Investigator — Service de Soins de Suites et Réadaptation Neurologique, Hôpital de la Pitié-Salpêtrière, 47/83 Bd de l'Hôpital, 75651 Paris Cedex 13
Locations (1):
- INSERM - Plateau IRM du CENIR, CR-ICM Hôpital Pitié-Salpêtrière, 47/83 Boulevard de l'Hôpital, Paris, Cedex 13, France